CLINICAL TRIAL: NCT02172690
Title: Laparoscopic Staging in Patients With Locally Advanced Gastric Cancer in Chinese Patients
Brief Title: Laparoscopic Staging for Locally Advanced Gastric Cancer in Chinese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jiafu Ji, Professor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KW-LStaging-2014; D141100000414004 (Other Grant/Funding Number: Beijing Municipal Science & Technology Commission)
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer; Peritoneal Metastases
Keywords: Gastric Cancer; Laparoscopic Staging; Cytology; Peritoneal Metastases
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laparoscopic Staging (Experimental): For Patients diagnosed as Locally Advanced Gastric Cancer(cT2+NanyM0)by CT and EUS, undergo laparoscopic staging.
  Interventions: Procedure: Laparoscopic Staging

INTERVENTIONS:
Procedure: Laparoscopic Staging — Laparoscopic Staging

SUMMARY:
RATIONALE: Laparoscopic staging may help doctors plan more effective treatment for gastric cancer, yet the efficiency have not been fully investigated in Chinese people.

PURPOSE: Study the effectiveness of laparoscopic staging in patients with pre-diagnosed as locally advanced gastric cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility of laparoscopic staging of patients with pre-diagnosed as locally advanced gastric cancer. II. Assess the adverse effects associated with this technique.

OUTLINE: Surgery. Laparoscopy with cytologic examination.

PROJECTED ACCRUAL: Up to 450 patients will be accrued over approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* sign written informed consent form
* age ≥ 18 years
* pathologically confirmed gastric or GEJ adenocarcinoma
* disease at clinical stage of locally advanced gastric cancer by CT/EUS(cT2+NanyM0)
* No prior antitumor treatment is allowed, including chemotherapy, radiotherapy, immune therapy or target therapy
* Adequate organ function as defined below:

Hematologic ANC ≥ 1.5*109/l Hemoglobin ≥ 9 g/dl Platelets ≥ 100*109/l Hepatic Albumin ≥ 30g/l Serum bilirubin ≤ 1.5×ULN AST and ALT ≤ 2.5×ULN ALP ≤ 2.5×ULN TBIL ≤ 1.5×ULN Renal Serum Creatinine < 1.5 ULN

* KPS ≥ 70
* Adequate lung and heart function
* Negative serum or urine pregnant test within 7 days prior to randomization for child-bearing age women
* Sexually active males or females willing to practice contraception during the study until 30 days after end of study.

Exclusion Criteria:

* Refuse to provide blood/tissue sample；
* With distant metastasis diagnosed by CT/EUS；
* Sexually active males or females refuse to practice contraception during the study until 30 days after end of study.
* History of organ transplantation（including autologous bone marrow transplantation and Peripheral stem cell transplantation）；
* Prior long term steroid therapy (excluding short term steroid treatment which is completed prior to > 2 weeks of study enrollment)；
* Patients with central nervous system(CNS) disorder or peripheral nervous system disorder or psychiatric disease；
* Concurrent severe infection；
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety (including current active hepatic, biliary, renal, respiratory disease, uncontrolled diabetes hypertension et al)；
* History of other malignancy. However, subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma, are eligible；
* Known history of uncontrolled or symptomatic angina, uncontrolled arrhythmias and hypertension, or congestive heart failure, or cardiac infarction within 6 months prior to study enrollment, or cardiac insufficiency；
* Person with no capacity (legally) or inappropriate to continue study treatment for ethics/medical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Peritoneal Metastasis or Positive Cytology | 7days

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 30days
  Number of Participants with Adverse Events(III or IV grades according to NCI-CTC)

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu Ji, MD, Principal Investigator — Peking University
Locations (1):
- Peking Unicersity Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li Z, Li Z, Zhang L, Liu Q, Wang Z, Zhang Z, Xiao G, Fu W, Wang X, Ye Y, Yu J, Li F, Chen L, Wang S, Ji J. Staging laparoscopy for locally advanced gastric cancer in Chinese patients: a multicenter prospective registry study. BMC Cancer. 2018 Jan 10;18(1):63. doi: 10.1186/s12885-017-3791-6. PMID 29321007